CLINICAL TRIAL: NCT05733689
Title: Response Adapted Neoadjuvant Therapy in Gastroesophageal Cancers (RANT-GC Trial) - a Phase Ib Feasibility Trial
Brief Title: Response Adapted Neoadjuvant Therapy in Gastroesophageal Cancers (RANT-GC Trial)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: BillionToOne, Inc (Unknown)
Responsible Party: Principal Investigator, Farshid Dayyani, Professor of Clinical Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1977; UCI 21-191 (Other: CFCCC)
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Gastroesophageal Adenocarcinoma
MeSH Terms: interventions — Folfox protocol; IFL protocol; folfirinox; Paclitaxel; Carboplatin; Docetaxel; Irinotecan; Single Person; Nivolumab; pembrolizumab; durvalumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant chemotherapy with ctDNA testing (Experimental): The patients will be treated with one of the standard neoadjuvant protocols (FLOT or FOLFOX.) If patient response to their treatment, as measured by CT Scans or MRI results or blood tests done to look tumor markers such as carcinoembryonic antigen (CEA) and Carbohydrate antigen 19-9 (CA19-9) a change in adjuvant treatment will be made.
  Interventions: Combination Product: FLOT; Combination Product: FOLFOX; Combination Product: FOLFIRI; Combination Product: FOLFIRINOX; Combination Product: PACLITAXEL with or without CARBOPLATIN; Combination Product: DOCETAXEL and IRINOTECAN (alone or combined); Drug: NIVOLUMAB (alone or when added to a regimen above); Drug: PEMBROLIZUMAB (alone or when added to a regimen above); Drug: Durvalumab; Drug: Trastuzumab

INTERVENTIONS:
Combination Product: FLOT — * Oxaliplatin 85 mg/m2 IV on Day 1
  * Docetaxel 50 mg/m2 IV on Day 1
  * Leucovorin 200 mg/m2 IV on Day 1
  * Fluorouracil 2600 mg/m2 continuous infusion over 24 hours daily on Day 1 Every 14 Days
Combination Product: FOLFOX — * Oxaliplatin 85 mg/m2 IV on Day 1
  * Leucovorin 400 mg/m2 IV on Day 1
  * Fluorouracil 400 mg/m2 IV Push on Day 1
  * Fluorouracil 1200 mg/m2 continuous infusion over 24 hours daily on Days 1 and 2 Every 14 Days
Combination Product: FOLFIRI — * Irinotecan 180 mg/m2 IV on Day 1
  * Leucovorin 400 mg/m2 IV on Day 1
  * Fluorouracil 400 mg/m2 IV Push on Day 1
  * Fluorouracil 1200 mg/m2 continuous infusion over 24 hours daily on Days 1 and 2 Every 14 Days
Combination Product: FOLFIRINOX — * Oxaliplatin 85 mg/m2 IV on Day 1
  * Irinotecan 150 mg/m2 IV on Day 1
  * Leucovorin 200 mg/m2 IV on Day 1
  * Fluorouracil 1200 mg/m2 continuous infusion over 24 hours daily on Days 1 and 2 Every 14 days
Combination Product: PACLITAXEL with or without CARBOPLATIN — * Paclitaxel 200 mg/m2 IV on Day 1
  * Carboplatin AUC 5 IV on day 1 Every 21 Days
  OR
  - Paclitaxel 80mg/m2 IV on Days 1,8,15 Every 28 Days
Combination Product: DOCETAXEL and IRINOTECAN (alone or combined) — * Docetaxel 35 mg/m2 IV on Days 1 and 8
  * Irinotecan 50 mg/m2 IV on Days 1 and 8 Every 21 Days
  * Docetaxel 75 mg/m2 IV on Day 1 Every 21 Days
  * Docetaxel 150 mg/m2 IV on Day 1 Every 14 Days
Drug: NIVOLUMAB (alone or when added to a regimen above) — * 240 mg IV on Day 1 every 14 days, or
  * 360 mg IV on Day 1 every 21 days, or
  * 480 mg IV on Day 1 every 28 days
Drug: PEMBROLIZUMAB (alone or when added to a regimen above) — * 200 mg IV on Day 1 every 21 days, or
  * 400 mg IV on Day 1 every 42 days
Drug: Durvalumab — - 1500 mg IV on Day 1 every 28 days
Drug: Trastuzumab — * 8 mg/kg on Day 1, then 6 mg/kg IV every 21 days, or
  * 6 mg/kg on Day 1, then 4 mg/kg IV every 14 days

SUMMARY:
This is a phase 1b prospective, single arm, open-label trial determining the efficacy and feasibility of using a response-guided approach to help guide neoadjuvant chemotherapy in subjects with Stage IB, II or Stage III adenocarcinoma of the stomach or gastroesophageal junction (GEA).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction (GEA). Other GE histologies which are treated per NCCN guidelines for neoadjuvant treatment are eligible.
* Must have Stage IB, II or Stage III GEA eligible for (neo)adjuvant doublet or triplet chemotherapy for up to 6 months.
* Age ≥ 18 years Because the safety or efficacy of neoadjuvant chemotherapy for LGEA has not been tested or established for patients <18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable.
* Performance status: ECOG performance status ≤2
* Life expectancy of greater than 6 months
* Adequate organ and marrow function as defined below:

  1. hemoglobin ≥ 7g/dL
  2. absolute neutrophil count ≥ 1,500/mcL
  3. platelets ≥ 80,000/mcl
  4. total bilirubin within normal institutional limits
  5. AST(SGOT)/ALT(SPGT) ≤ 5 X institutional upper limit of normal
  6. creatinine <2 X ULN
* Docetaxel can cause fetal harm and irinotecan is known to be teratogenic. Since these compounds are part of the treatment regimens, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  1. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  1. Has not undergone a hysterectomy or bilateral oophorectomy; or
  2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent. 1. Both men and women and members of all races and ethnic groups are eligible for this trial. Non-English speaking, deaf, hard of hearing and illiterate individuals are eligible for this trial.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients with known distant metastases from GEA.
* History of allergic reactions attributed to agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of another primary cancer which requires active treatment or is expected to require treatment within 12 months after enrollment.
* Inability to comply with study and follow-up procedures as judged by the Investigator.
* Patients who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Patients with prior organ/bone marrow/non-autologous stem cell transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of completing per protocol treatment. | Up to 3 years
  Percent of patients who will undergo attempt at curative intent resection.

SECONDARY OUTCOMES:
Percentage of patients completing gastrectomy. | Up to 3 years
  Percent of patients completing gastrectomy
Rate of negative ctDNA after completion of neoadjuvant treatment and within 8 weeks after surgery | 8 weeks
  Percent of patients with ctDNA clearance after neoadjuvant chemotherapy and after surgery (within 6-8 weeks)
Rate of R0 resection | Up to 3 years
  R0 resection is defined as complete tumor removal with negative surgical margins.
Percentage of Grade 3-5 Adverse Events | Up to 3 years
  Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.
Relapse-free survival time | Up to 3 years
  The lead time in ctDNA detection before clinical recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Dayyani, MD,PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No